CLINICAL TRIAL: NCT01131572
Title: N-acetylcysteine in Bulimia Nervosa
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB19223, 09-09-18-01
Record Dates: First submitted 2010-05-24; First posted 2010-05-27 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: NAC
MeSH Terms: interventions — Acetylcysteine

ARMS (1):
- N-acetylcysteine (Other): open label treatment. Each subject receives N-acetylcysteine.
  Interventions: Drug: N-acetylcysteine NAC

INTERVENTIONS:
Drug: N-acetylcysteine NAC — N-acetylcysteine in the treatment of Bulimia Nervosa

SUMMARY:
This study tests NAC in the treatment of Bulimia Nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Bulimia Nervosa
* 18-65 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Binge-purge episodes | per week
  The primary outcome measure will be the weekly frequency of binge-purge episodes. A binge-purge eating episode will be defined using DSM-IV-TR criteria, and accessed via clinical interview and review of subject take-home diaries at each study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

REFERENCES:
- [Result] Guerdjikova AI, Blom TJ, Mori N, McElroy SL. N-acetylcysteine in bulimia nervosa--open-label trial. Eat Behav. 2013 Jan;14(1):87-9. doi: 10.1016/j.eatbeh.2012.11.001. Epub 2012 Nov 19. PMID 23265409
- See also: Lindner Center of HOPE research page — http://lindnercenterofhope.org/research